CLINICAL TRIAL: NCT01825408
Title: A Randomized Cohort Trial Evaluating Duration of Antibiotic Therapy as Part of Maximal Medical Therapy for Chronic Rhinosinusitis
Brief Title: Duration of Antibiotic Therapy as Part of Maximal Medical Therapy for Chronic Rhinosinusitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Adam Zanation, MD, Assistant Professor of Otolaryngology/Head and Neck Surgery, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-2377
Record Dates: First submitted 2013-03-18; First posted 2013-04-05 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Sinusitis
MeSH Terms: conditions — Sinusitis | interventions — Doxycycline; Azithromycin; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Doxycycline, 3 weeks (Active Comparator): Subjects with chronic rhinosinusitis with nasal polyps (CRSwNP) will receive Doxycycline 100mg BID or if allergic to doxycycline, then Augmentin 875mg BID for 3 weeks duration. These patients will also receive a course of Prednisone (30mg x 3d, 20mg x 3d, 10mg x3d, 10mg every other day for 6 days (3 doses)) which is standard of care treatment for patients with chronic sinusitis with nasal polyps.
  Interventions: Drug: Doxycycline; Drug: Augmentin
- Doxycycline, 6 weeks (Active Comparator): Subjects with Chronic Rhinosinusitis with Nasal Polyps (CRSwNP)will receive Doxycycline 100mg BID or if allergic to doxycycline, then Augmentin 875mg BID for 6 weeks duration. These patients will also receive a course of Prednisone (30mg x 3d, 20mg x 3d, 10mg x3d, 10mg every other day for 6 days (3 doses)) which is standard of care treatment for patients with chronic sinusitis with nasal polyps.
  Interventions: Drug: Doxycycline; Drug: Augmentin
- Azithromycin, 3 weeks (Active Comparator): Subjects with Chronic Rhinosinusitis without Nasal Polyps will receive Azithromycin 250mg daily, or if allergic to azithromycin, then Augmentin 875mg BID for 3 weeks duration.
  Interventions: Drug: Azithromycin; Drug: Augmentin
- Azithromycin, 6 weeks (Active Comparator): Subjects with chronic Rhinosinusitis without Nasal Polyps will receive Azithromycin 250mg daily, or if allergic to azithromycin, then Augmentin 875mg BID for 6 weeks duration.
  Interventions: Drug: Azithromycin; Drug: Augmentin

INTERVENTIONS:
Drug: Doxycycline — Subjects with CRSwNP who are not allergic to doxycycline will receive Doxycycline 100mg BID for either 3 or 6 weeks duration.
  Arms: Doxycycline, 3 weeks; Doxycycline, 6 weeks
Drug: Azithromycin — Subjects with CRS without Nasal Polyposis (CRSwNP)who are not allergic to azithromycin will be given Azithromycin 250mg daily for either 3 or 6 weeks duration.
  Arms: Azithromycin, 3 weeks; Azithromycin, 6 weeks
Drug: Augmentin — If a subject in any of the study arms is allergic to the medication he/she is supposed to receive, he/she will be given Augmentin 875mg BID for either 3 or 6 weeks duration

SUMMARY:
The purpose of this study is to determine the best duration(3 versus 6 weeks) of antibiotics as part of maximal medical therapy for treating chronic sinusitis and thus preventing patients from having to have sinus surgery. The hypothesis is that in the context of maximal medical therapy 3 weeks of antibiotics is not worse than 6 weeks of antibiotics at successfully treating chronic sinusitis.

DETAILED DESCRIPTION:
OVERVIEW This is a prospective randomized cohort study assessing duration of antibiotics (3 vs 6 weeks) as part of maximal medical therapy for chronic rhinosinusitis. Up to 100 subjects will be prospectively enrolled from patients visiting the Department of Otolaryngology-Head and Neck Surgery clinics at UNC Hospitals.

INITIAL CLINIC VISIT At the time of a clinical visit, the attending otolaryngologists will identify their patients with chronic rhinosinusitis (CRS) who are appropriate for maximal medical treatment, including antibiotics. They will introduce the study to these patients and invite them to learn more about it.

If the patient is interested in learning more about the study, the study coordinators will be contacted to provide additional information and, if the patient would like to participate in the study, provide informed consent.

If the patient is a premenopausal woman, she will be asked if she is pregnant or breastfeeding.

If she is either of these, she will be excluded from the study. All remaining women will receive a urine pregnancy test. If this urine pregnancy test is positive, the patient will be excluded from the study. Thus, for premenopausal female patients, a negative urine pregnancy test is necessary for inclusion in the study. These women will be informed that they should use an effective method of birth control during the study:

* Combined oral contraceptives
* Patch contraceptives
* Vaginal ring contraceptives
* Injectable contraceptives
* Implantable contraceptives
* Intrauterine devices or intrauterine systems
* Tubal ligation
* Barrier methods of contraception (male condom, female condom, cervical cap with spermicide, or diaphragm with spermicide)
* Vasectomy of your partner in a monogamous relationship

Women enrolled in this study will be informed that if they have a failure of birth control method during the course of the study or become pregnant during the study, they will be withdrawn from the study and further treatment will be decided according to the clinical withdrawn from the study and further treatment will be decided according to the clinical expertise of the treating otolaryngologist.

* The study coordinators will assign the patients a unique Subject ID that will be used on all patient forms with the exception of the informed consent documents and HIPAA authorization forms.
* The patient will fill out a demographics and past medical history form.
* Using a random-number generator, the patient will be randomized to receive either 3 or 6 weeks of antibiotics.
* The subject will initially be given a prescription for empiric antibiotics.The choice of empiric antibiotics will differ based on the patient's nasal polyposis status:
* If the subject has CRS with nasal polyposis (CRSwNP), s/he will be given Doxycycline 100mg BID or if allergic to doxycycline, then Augmentin 875mg BID for either 3 or 6 weeks duration. These patients will also receive a course of Prednisone (30mg x 3d, 20mg x 3d, 10mg x3d, 10mg every other day for 6 days (3 doses)) which is standard of care treatment for CRSwNP.
* If the subject has CRS without Nasal Polyposis (CRSwNP), s/he will be given Azithromycin 250mg daily, or if allergic to azithromycin, then Augmentin 875mg BID for either 3 or 6 weeks duration.
* If purulent nasal discharge is present that is appropriate for culture, the otolaryngologists will send this for culture and sensitivity analysis, which they would normally do as part of their routine clinical care. The patients will be informed that if their culture and sensitivity analysis indicates that they have an infection that can be treated with a less broad-spectrum antibiotic, then they will be prescribed culture-directed antibiotics. Otherwise, the patient can continue empiric antibiotics as previously specified.
* All study participants will also be prescribed standard of care intranasal steroids, and encouraged to perform BID saline sinus irrigation and use yogurt/over the counter probiotics to reduce GI side effects of antibiotics.

4-5 WEEKS AFTER BEGINNING TREATMENT For subjects randomized to the 3 week antibiotic group, these subjects will been seen in clinic.

During this visit (study visit #2), subjects will be asked about antibiotic compliance and side effects. Recommendation for sinus surgery will be evaluated with video-recorded nasal endoscopy and a sinus CT and made based on clinical judgement.

For subjects randomized to the 6 week antibiotic group, these subjects will be contacted by phone by the study coordinator to assess side effects and medication compliance.

7-8 WEEKS AFTER BEGINNING TREATMENT

For subjects randomized to the 6 week antibiotic group, these subjects will been seen in clinic.

During this visit (study visit #2), subjects will be asked about antibiotic compliance and side effects. Recommendation for sinus surgery will be evaluated with video-recorded nasal endoscopy and a sinus CT and made based on clinical judgement.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic rhinosinusitis
* 18 years of age or older
* English speaking

Exclusion Criteria:

* Pregnant or breastfeeding women
* vasculitis
* cystic fibrosis
* primary ciliary dyskinesia
* allergic fungal sinusitis
* gross immunodeficiency
* current use of chemotherapy
* insulin-dependent diabetes mellitus
* recent trial of maximal medical therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Zanation, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Department of Otolaryngology-Head and Neck Surgery clinics at UNC Hospitals, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Doxycycline, 3 Weeks | Doxycycline, 6 Weeks | Azithromycin, 3 Weeks | Azithromycin, 6 Weeks
Started | 7 | 7 | 14 | 12
Completed | 7 | 7 | 14 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxycycline, 3 Weeks | Doxycycline, 6 Weeks | Azithromycin, 3 Weeks | Azithromycin, 6 Weeks | Total
Number analyzed (Participants) | 7 | 7 | 14 | 12 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 11 | 9 | 33
  >=65 years | 1 | 0 | 3 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 8 | 8 | 21
  Male | 4 | 5 | 6 | 4 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Recommended for Sinus Surgery After 3 Weeks of Antibiotic Therapy
Description: Recommendation for sinus surgery after completion of maximal medical therapy is determined by the subject's treating physician and is based on two citeria: (1) persistence of symptoms and (2) objective evidence of disease on post-treatment sinus CT scan or nasal endoscopy. Symptomatic improvement of sinusitis symptoms will be assessed by: patient self report, change in Chronic Sinusitis Survery (CSS) score and change in RhinoSinusitis Disibility Index (RSDI) score relative to initial pre-antibiotic CSS and RSDI survey scores.
Time Frame: 4-5 weeks after starting antibiotics
Measure: Count of Participants; unit: Participants
Arm/Group | Doxycycline, 3 Weeks | Azithromycin, 3 Weeks
Number analyzed (Participants) | 7 | 14
Participants
  Sinus Surgery Recommended | 7 | 8
  Sinus Surgery NOT Recommended | 0 | 6

2. Primary Outcome: Number of Patients Recommended for Sinus Surgery After 6 Weeks of Antibiotic Therapy
Description: as for outcome 1
Time Frame: 7-8 weeks after initiating antibiotics
Measure: Count of Participants; unit: Participants
Arm/Group | Doxycycline, 6 Weeks | Azithromycin, 6 Weeks
Number analyzed (Participants) | 7 | 12
Participants
  Sinus Surgery Recommended | 5 | 8
  Sinus Surgery NOT Recommended | 2 | 4

ADVERSE EVENTS:
Arm/Group | Doxycycline, 3 Weeks | Doxycycline, 6 Weeks | Azithromycin, 3 Weeks | Azithromycin, 6 Weeks
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 0/7 | 1/7 | 0/14 | 1/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Doxycycline, 3 Weeks (N=7) | Doxycycline, 6 Weeks (N=7) | Azithromycin, 3 Weeks (N=14) | Azithromycin, 6 Weeks (N=12)
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No